CLINICAL TRIAL: NCT06764940
Title: A Pivotal Phase II Clinical Trial of Utidelone Injection (UTD1) Plus Capecitabine (CAP) in HER2-negative Breast Cancer Patients With Brain Metastases
Brief Title: A Pivotal Phase II Clinical Trial of Utidelone Injection Plus Capecitabine in HER2-negative Breast Cancer Patients With Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biostar Pharma, Inc. (Industry)
Responsible Party: Sponsor
Organization: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG01-2402
Record Dates: First submitted 2025-01-07; First posted 2025-01-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: HER2-negative Breast Cancer Patients With Brain Metastases
Keywords: breast cancer; brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- (stage 1) monotherapy group (Experimental)
  Interventions: Drug: Utidelone
- (stage 1) combination group A (Experimental)
  Interventions: Drug: Utidelone in combination with capecitabine
- (stage 1) combination group B (Experimental)
  Interventions: Drug: Utidelone in combination with capecitabine
- (stage 2) combination group (Experimental)

INTERVENTIONS:
Drug: Utidelone — Utidelone 30 mg/m2/d i.v, once a day for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: (stage 1) monotherapy group
Drug: Utidelone in combination with capecitabine — UTD1 25 mg/m2/d i.v, once a day for 5 consecutive days, every 21 days as a treatment cycle plus capecitabine 1000 mg/m2 orally twice a day, for 1 to 14 days, 21 days as a treatment cycle.
  Arms: (stage 1) combination group B
Drug: Utidelone in combination with capecitabine — Utidelone 30 mg/m2/d i.v, once a day for 5 consecutive days, every 21 days as a treatment cycle plus capecitabine 1000 mg/m2 orally twice a day, for 1 to 14 days, 21 days as a treatment cycle.
  Arms: (stage 1) combination group A
Drug: Utidelone in combination with capecitabine — Utidelone 25 mg/m2/d or 30 mg/m2/d i.v, once a day for 5 consecutive days, every 21 days as a treatment cycle plus capecitabine 1000 mg/m2 orally twice a day, for 1 to 14 days, 21 days as a treatment cycle.

SUMMARY:
This study is a multicenter, two-stage clinical trial to evaluate the efficacy and safety of utidelone in combination with capecitabine in patients with HER2-negative breast cancer with brain metastases. Patients will be enrolled to receive treatment of utidelone alone or in combination with capecitabine.

The objectives both in stage I and stage II are to evaluate the intracranial and systemic efficacy and safety of utdelone plus capecitabine for the treatment of HER2-negative breast cancer patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed HER2-negative metastatic breast cancer. HER2-negative defined as immunohistochemical (IHC) score of 0 or 1+, or IHC2+ with negative HER2 expression on in situ hybridization (ISH).
2. Based on screening contrast-enhanced brain MRI, patients must have at least one measurable intracranial lesion according to RECIST 1.1 (≥1.0 cm in size) .
3. Male or female aged ≥18 years.
4. ECOG PS 0 or 1.
5. Have a life expectancy of at least 3 months.
6. Have adequate baseline hematologic parameters.
7. Have adequate hepatic and renal function.
8. ≤ 3 prior lines of chemotherapy in advanced or metastatic setting.
9. Women of childbearing potential, unless hysterectomy or oophorectomy or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to study drug administration] sexual partner) for at least 4 weeks prior to study drug administration, during study and up to 6 months following the last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician. Investigator will discuss with patient on the above points and the patient agreement will be documented in the source document. The investigator should ensure that the patient is using an effective method of avoiding pregnancy as per protocol. In case of Male patients: Either patient partners or patients themselves must use an effective method of avoiding pregnancy for at least 4 weeks prior to study drug administration, during study and up to 6 months following the last dose.
10. Patients must be able to follow the study visit schedule, and must be able of sign and give informed consent in accordance with institutional review board.

Exclusion Criteria:

1. Leptomeningeal metastasis confirmed by MRI and/or cerebrospinal fluid cytology.
2. Any intracranial lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to patient (e.g. brain stem lesions).
3. Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy.
4. Had evidence of intracranial hemorrhage within 3 months before study treatment.
5. Had evidence of hemoptysis within 6 months before study treatment. Or bleeding or evidence of coagulopathy within 4 weeks before study treatment.
6. Undergone major surgical procedures within 4 weeks or not fully recovered from surgery before study treatment.
7. Patients who have received anti-tumor therapies less than 2 weeks before the first dose of investigational product, including endocrine therapy, chemotherapy, radiotherapy, biotherapy, targeted therapy, immunotherapy or antibody-drug conjugate therapy.
8. Persistent toxicities caused by previous antitumor therapy (excluding alopecia), not yet improved to CTCAE v5.0 grade ≤ 1 or baseline.
9. Patients with neuropathy> grade 1.
10. Known hypersensitivity to any components of the investigational product.
11. Known deficiency of dihydropyrimidine dehydrogenase (DPD).
12. This applies only to the combination cohort and does not apply to the monotherapy cohort. For patients with previous capecitabine treatment, the prior use of capecitabine meets any of the following criteria: A) The best response during prior capecitabine combination therapy or monotherapy is Progressive Disease (PD); B) Have received capecitabine treatment within 6 months prior to the first study treatment.
13. Patients who are pregnant (positive pregnancy test) or lactating.
14. Patients with other malignancies over the past 5 years, except for inactive tumors with good prognosis, including resected basal cell and squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, or papillary thyroid cancer.
15. Patients who are particpating in other interventional studies or who are receiving other study treatments (patients who have discontinued other investigational treatments and are in follow-up are eligible for enrollement in this study).
16. Known active or uncontrolled hepatitis B infection, active syphilis, or HIV infection that is not well controlled; or positive for hepatitis B virus based on the evaluation of results of tests for hepatitis B (HBsAg, anti-HBs, anti-HBc, or HBV DNA) infection at screening.
17. With a history of severe or uncontrolled diseases.
18. Autoimmune diseases requiring treatment with systemic glucocorticoids.
19. Not able to perform contrast-enhanced brain MRI or known contraindications to MRI gadolinium contrast, such as cardiac pacemaker, shrapnel, or eye foreign body.
20. Patients with a history of other systemic severe diseases or abnormal laboratory findings that would, in the Investigator's judgment, be inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective Response Rate (IC-ORR) evaluated by investigator according to RECIST 1.1 criteria. | 12 months

SECONDARY OUTCOMES:
IC-ORR evaluated by investigator according to Neuro-Oncology Brain Metastases criteria (RANO-BM). | 12 months
ORR according to RECIST 1.1 criteria. | 12 months
Progression Free Survival (PFS) according to RECIST 1.1 criteria. | 12 months
Disease Control Rate (DCR) according to RECIST 1.1 criteria. | 12 months
Duration of Response (DOR) according to RECIST 1.1 criteria. | 12 months
Intracranial Progression Free Survival (IC-PFS) according to RECIST 1.1 criteria and RANO-BM. | 12 months
Intracranial Disease Control Rate (IC-DCR) according to RECIST 1.1 criteria and RANO-BM. | 12 months
Intracranial Duration of Response (IC-DOR) according to RECIST 1.1 criteria and RANO-BM. | 12 months
Overall Survival (OS) | up tp 24 months
Treatment-emergent Adverse Event-TEAE | Until 28 days after the last dose of treatment

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - City of Hope--Duarte, Duarte, California
  - Cancer & Blood Research Center, LLC, Los Alamitos, California
  - Univ. of California Los Angeles, Los Angeles, California
  - FOMAT Medical Research (Network), Oxnard, California
  - Scripps Health, San Diego, California
  - University Of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Biosresearch Partner, Hialeah, Florida
  - D&H Cancer Research Center, Margate, Florida
  - Augusta University, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center Northwestern University, Chicago, Illinois
  - The Johns Hopkins Sidney Kimmel Cancer Center, Johns Hopkins School of Medicine, Baltimore, Maryland
  - Profound Research LLC, Farmington Hills, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Stony Brook Cancer Center, Stony Brook, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Community Clinical Trials, Kingwood, Texas
  - Tranquil Clinical Research, Webster, Texas

IPD SHARING:
Plan to Share IPD: No